CLINICAL TRIAL: NCT05855408
Title: Effectiveness of a Second COVID-19 Vaccine Booster in Chinese Adults Aged 18 Years or Above: a Multicenter, Parallel Groups, Partially Randomized, Open-label, Blank-controlled Adaptive Platform Trial
Brief Title: Effectiveness of a Second COVID-19 Vaccine Booster in Chinese Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT178
Record Dates: First submitted 2023-05-10; First posted 2023-05-11 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; effectiveness; hybrid immunity; booster immunization; adaptive platform trial
MeSH Terms: conditions — COVID-19 | interventions — SYS6006 COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Subjects are assigned to receive one dose of intramuscularly administered Ad5-nCoV vaccine as the second booster.
  Interventions: Biological: Intramuscularly administered Ad5-nCoV vaccine
- Group 2 (Experimental): Subjects are assigned to receive one dose of aerosolized Ad5-nCoV vaccine as the second booster.
  Interventions: Biological: Aerosolized Ad5-nCoV
- Group 3 (Experimental): Subjects are assigned to receive two doses of DelNS1-2019-nCoV-RBD-OPT1 vaccine as the second booster.
  Interventions: Biological: DelNS1-2019-nCoV-RBD-OPT1
- Group 4 (Experimental): Subjects are assigned to receive one dose of SYS6006 vaccine as the second booster.
  Interventions: Biological: SYS6006
- Group 5 (No Intervention): Subjects are not assigned any vaccines served as a blank control.

INTERVENTIONS:
Biological: Intramuscularly administered Ad5-nCoV vaccine — This vaccine is produced by CanSino Biologics Inc.
  Arms: Group 1
Biological: Aerosolized Ad5-nCoV — This vaccine is produced by CanSino Biologics Inc.
  Arms: Group 2
Biological: DelNS1-2019-nCoV-RBD-OPT1 — This vaccine is produced by Wantai Biopharmaceutical Company.
  Arms: Group 3
Biological: SYS6006 — This vaccine is produced by CSPC Pharmaceutical Group Co., Ltd.
  Arms: Group 4

SUMMARY:
This is a multicenter, parallel groups, partially randomized, open-label, blank-controlled adaptive platform study to evaluate the effectiveness of a second COVID-19 vaccine booster in Chinese adults who are charactered as the majority of whom with hybrid immunity of COVID-19 vaccination and COVID-19 breakthrough infection. Individuals aged 18 years and over, include the elderly over 60 years old or those with underlying diseases (history of underlying medical conditions diagnosed by a clinician, including hypertension, diabetes, heart disease, etc). The eligible participants with an interval ≥ 4 months after previous SARS-CoV-2 infection (or had never been infected) and ≥ 6 months from the first COVID-19 vaccine booster will be recruited. Participants who are not willing to receive the second booster but are consent to participate the surveillance for COVID-19, will be included as a blank control. Informed consent will be acquired from eligible participants. Other participants who are willing to receive the second booster and participate the surveillance for COVID-19, will be randomly allocated in a ratio of 1: k (k is the number of vaccine types) to the different investigational vaccines, stratified according to age and history of COVID-19 infection. The symptomatic COVID-19 cases will be reported and documented in both the investigational and control groups. The occurrence of serious adverse events within 6 months after vaccination will be observed. Moreover, blood and nasal mucosa samples will be collected on the day 0 before and day 14, month 3 and 6 after the booster vaccination in a subgroup for humoral, cellular and mucosal immunogenicity analysis. Moreover, oral specimens will be collected once for all participants on the day of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and over, including the elderly over 60 years and those with underlying diseases.
2. Volunteers are able and willing to comply with the requirements of the clinical trial protocol and sign the informed consent form.
3. ≥ 4 months from the last SARS-CoV-2 infection (or never been infected), and 6 months or more from the first booster immunization of the COVID-19 vaccine.

Exclusion Criteria:

1. Volunteers have suspected symptoms of COVID-19 when enrolled, such as dry throat, sore throat, cough, etc.
2. The COVID-19 Antigen Quick Test Kit is positive when volunteers are enrolled.
3. Fever, temperature > 37.0°C.
4. Have received a second COVID-19 vaccine booster immunization.
5. Have a history of serious adverse reactions related to the vaccine and/or have a history of severe allergic reactions to any component of the investigational vaccine (only applicable to the vaccine groups).
6. Pregnant or lactating women.
7. HIV infection, tuberculosis, low immunity caused by disease or long-term medication.
8. Acute disease or acute onset of chronic disease.
9. Epilepsy and other progressive neurological disorders.
10. Other situations that are not suitable for participating in this research, according to the judgment of the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-18 (Estimated); Primary Completion 2024-05-18 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of COVID-19 from 14 days to 6 months after the booster immunization. | from 14 days to 6 months after the booster dose

SECONDARY OUTCOMES:
The incidence of COVID-19 from 7 days to 6 months after the booster immunization. | from 7 days to 6 months the booster dose
The incidence of COVID-19 from 28 days to 6 months after the booster immunization. | from 28 days to 6 months the booster dose
The incidence of graded COVID-19 (mild, moderate, severe, critical or death) from 7 days to 6 months after the booster immunization. | from 7 days to 6 months the booster dose
The incidence of graded COVID-19 (mild, moderate, severe, critical or death) from 14 days to 6 months after the booster immunization. | from 14 days to 6 months the booster dose
The incidence of graded COVID-19 (mild, moderate, severe, critical or death) from 28 days to 6 months after the booster immunization. | from 28 days to 6 months the booster dose
The incidence of hospitalized COVID-19 from 7 days to 6 months after the booster immunization. | from 7 days to 6 months the booster dose
The incidence of hospitalized COVID-19 from 14 days to 6 months after the booster immunization. | from 14 days to 6 months the booster dose
The incidence of hospitalized COVID-19 from 28 days to 6 months after the booster immunization. | from 28 days to 6 months the booster dose
Geometric mean titer (GMT), Geometric mean fold increase (GMFI) and seroconversion of neutralizing antibodies against wild-type SARS-CoV-2 and omicron variant on day 14 after the booster vaccination in the immunogenic subgroup. | On day 14 after the booster vaccination
GMT, GMFI and seroconversion of neutralizing antibodies against wild-type SARS-CoV-2 and omicron variant on month 3 after the booster vaccination in the immunogenic subgroup. | On month 3 after the booster vaccination
GMT, GMFI and seroconversion of neutralizing antibodies against wild-type SARS-CoV-2 and omicron variant on month 6 after the booster vaccination in the immunogenic subgroup. | On month 6 after the booster vaccination
GMT, GMFI and seroconversion of S-RBD-specific IgG antibodies against wild-type SARS-CoV-2 and omicron variant on day 14 after the booster vaccination in the immunogenic subgroup. | On day 14 after the booster vaccination
GMT, GMFI and seroconversion of S-RBD-specific IgG antibodies against wild-type SARS-CoV-2 and omicron variant on month 3 after the booster vaccination in the immunogenic subgroup. | On month 3 after the booster vaccination
GMT, GMFI and seroconversion of S-RBD-specific IgG antibodies against wild-type SARS-CoV-2 and omicron variant on month 6 after the booster vaccination in the immunogenic subgroup. | On month 6 after the booster vaccination
GMT, GMFI and seroconversion of nasal specific IgA antibodies on day 14 after the booster vaccination in the immunogenic subgroup. | On day 14 after the booster vaccination
GMT, GMFI and seroconversion of nasal specific IgA antibodies on month 3 after the booster vaccination in the immunogenic subgroup. | On month 3 after the booster vaccination
GMT, GMFI and seroconversion of nasal specific IgA antibodies on month 6 after the booster vaccination in the immunogenic subgroup. | On month 6 after the booster vaccination
The incidence of serious adverse events within 6 months after the booster vaccination. | within 6 months after the booster dose

OTHER OUTCOMES:
The effectiveness for preventing COVID-19 from 7 days after the booster dose will be analyzed stratified based on the S-RBD IgG antibody level at enrollment. | on day 7 after the booster dose
The effectiveness for preventing COVID-19 from 14 days after the booster dose will be analyzed stratified based on the S-RBD IgG antibody level at enrollment. | on day 14 after the booster dose
The effectiveness for preventing COVID-19 on day 28 after the booster dose will be analyzed stratified based on the S-RBD IgG antibody level at enrollment. | on day 28 after the booster dose
Cross-neutralizing antibody levels against other variants on day 14 after the booster vaccination in the immunogenic subgroup. | On day 14 after the booster vaccination
Cross-neutralizing antibody levels against other variants on month 3 after the booster vaccination in the immunogenic subgroup. | On month 3 after the booster vaccination
Cross-neutralizing antibody levels against other variants on month 6 after the booster vaccination in the immunogenic subgroup. | On month 6 after the booster vaccination
Effectiveness and immunogenicity after the second booster immunization will be subgroup analyzed in the elderly over 60 years old and those with underlying diseases. | from 14 days to 6 months after the booster dose
The impact of the human genome on the effect of vaccination. | from 14 days to 6 months after the booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China